CLINICAL TRIAL: NCT02526329
Title: A Phase 1 Single Center Safety and Feasibility Study of Primary T Regulatory Cell Therapy to Treat Visceral Acute Graft-versus-Host Disease Following Hematopoietic Cell Transplantation
Brief Title: Donor Regulatory T Cells in Treating Patients With Visceral Acute Graft-versus-Host Disease After Stem Cell Transplant
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Logistics
Sponsor: Everett Meyer (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Everett Meyer, Assistant Professor of Medicine, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-30861; NCI-2014-01609 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB-30861 (Other: Stanford IRB); BMT267 (Other: OnCore)
Record Dates: First submitted 2015-08-14; First posted 2015-08-18 (Estimated); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Graft Versus Host Disease
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (donor regulatory T lymphocytes) (Experimental): Patients receive donor regulatory T lymphocytes intravenously (IV) over 5 minutes or less on day 0. Some patients receive a second infusion of frozen donor regulatory T lymphocytes 5-7 days after the initial infusion or 2 additional infusions separated by 5-7 days.
  Interventions: Biological: donor regulatory T lymphocytes; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: donor regulatory T lymphocytes — Given IV
  Other Names: donor CD4+CD25+FoxP3+ T cells
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of donor regulatory T cells in treating patients with graft-versus-host disease affecting the liver or gastrointestinal organs (visceral) within 100 days (acute) after undergoing a stem cell transplant. Graft-versus-host disease occurs when donor immune cells infused in a stem cell transplant attack the gut, skin, liver, or other organ systems of the patient. Regulatory T cells are a type of immune cell that may be able to reduce the attack of the donor's immune cells on the patient's normal cells and help treat graft-vs-host disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the safety and feasibility of donor T regulatory (Treg) cell infusions in subjects with visceral acute graft-versus-host disease (aGVHD) and incidence of dose limiting toxicities (DLTs) graded according to the Common Terminology Criteria for Adverse Events (CTCAE version 4 [v.4]) with a focus on infusion reactions within 24 hours, respiratory distress within 72 hours of infusion and all-cause mortality within 28 days of infusion.

SECONDARY OBJECTIVES:

I. Determine the quantitative blood Treg cell changes following the cell infusions.

II. Assess dosing requirements and treatment response rates to primary steroid, secondary and tertiary immunosuppressive therapy.

III. Post-transplant day +100 and day +180 survival. IV. Post-transplant incidence of chronic graft-versus-host disease (GVHD) at day +180.

OUTLINE: This is a dose-escalation study.

Patients receive donor regulatory T lymphocytes intravenously (IV) over 5 minutes or less on day 0. Some patients receive a second infusion of frozen donor regulatory T lymphocytes 5-7 days after the initial infusion or 2 additional infusions separated by 5-7 days.

After completion of study treatment, patients are followed up weekly until day 28 and then on days 100 and 180.

ELIGIBILITY:
Inclusion Criteria:

* Visceral aGVHD defined as: at least stage III/IV acute liver or stage II/III gastrointestinal (GI) GVHD by clinical criteria and/or GI and/or liver biopsy confirmation showing no alternative explanation for symptoms of GVHD
* Ability to understand and willingness to sign a written informed consent form
* Must have a 7/8 or 8/8 or haploidentical related donor matched at the human leukocyte antigen (HLA)-A, B, C, DRB1 who was evaluated and provided the donor transplant graft
* Myeloablative or non-myeloablative allogeneic hematopoietic cell transplantation
* Karnofsky performance status >= 50
* DONOR: Age >= 18 to =< 77 years old
* DONOR: Karnofsky performance status of >= 70% defined by institutional standards
* DONOR: Must be the same sibling donor from whom the recipient's blood and marrow graft was collected for the original allogeneic transplant that is HLA 7/8 or 8/8 or haploidentical matched at the HLA-A, B, C, and DRB1
* DONOR: Serologies for human immunodeficiency virus (HIV) antigen (Ag), HIV 1 and HIV 2 antibody (Ab), human T-cell lymphotropic virus (HTLV) 1 and HTLV 2 Ab, hepatitis B surface antigen (sAg) or polymerase chain reaction (PCR)+, or hepatitis C Ab or PCR+, syphilis (Treponema) screen and HIV 1 and hepatitis C by NAT (nucleic acid testing) have been collected prior to apheresis
* DONOR: Female donors of child-bearing potential must have a negative serum or urine beta-human chorionic gonadotropin (HCG) test within two weeks of apheresis
* DONOR: Capable of undergoing leukapheresis, have adequate venous access, and be willing to undergo insertion of a central catheter should leukapheresis via peripheral vein be inadequate
* DONOR: Donor selection will be in compliance with 21 Code of Federal Regulations (CFR) 1271

Exclusion Criteria:

* Uncontrolled infections not responsive to antimicrobial therapy requiring intensive critical care
* Progressive malignant disease, including post-transplant lymphoproliferative disease unresponsive to therapy
* Cytomegalovirus colitis or enteritis as defined by cytomegalovirus (CMV) shell vial or culture positivity from endoscopic biopsy the discretion of the treating physician based upon PCR positivity, clinical presentation and histology
* Respiratory insufficiency with oxygen requirement > 4 L nasal cannula
* Multi-organ failure
* DONOR: Evidence of active infection or viral hepatitis
* DONOR: HIV positive
* DONOR: Pregnant donor
* DONOR: Factors which place the donor at increased risk for complications from leukapheresis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-08-06 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade 3 infusion reaction within 24 hours of infusion | 24 hours
  Dose-limiting toxicity will be defined as CTCAE Grade 3 or higher cytokine/release syndrome/acute infusion reaction within 24 hours after Treg cell infusion. The rates of defined DLTs will be calculated and the one-sided upper 80%, 90%, and 95% confidence limits calculated.

SECONDARY OUTCOMES:
Incidence of grade 3 or higher non-GVHD infusion-related adverse events | Up to day 28
  Incidence of grade 3 or higher non-GVHD infusion-related adverse events according to the CTCAE v4 that are not anticipated following HCT will be reported
Grade 4 (life threatening) or 5 (fatal) adverse events | 28 days
  Grade 4 (life threatening) or 5 (fatal) adverse events within after 28 days of Treg infusion that were otherwise unexpected in the immediate post transplant setting will be reported
Grade 4 (life threatening) respiratory distress | 72 hours
  Grade 4 (life threatening) respiratory distress within 72 hours of Treg infusion will be reported
Change in blood Treg cell numbers following the infusions | Baseline to up to day 28
  The change in Treg cell counts from baseline to post infusion will be depicted in boxplots of both relative proportion and absolute numbers. Mean log (fold change) and confidence intervals will be calculated. The confidence intervals will be used to test the hypotheses of no change from baseline to post infusion.
Overall survival (OS) | Day 100
  The OS will be estimated by the Kaplan-Meier product-limit method, with standard confidence limits.
Incidence of cGVHD. | 180 days
  Incidence of cGVHD will be reported at Post HCT day +180

CONTACTS AND LOCATIONS:
Overall Officials: Everett Meyer, Principal Investigator — Stanford University Hospitals and Clinics
Locations (1):
- Stanford University Hospitals and Clinics, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No